CLINICAL TRIAL: NCT06273683
Title: Comparison of Two Salpingectomy Techniques for Sterilization at the Time of Cesarean Delivery
Status: Recruiting | Type: Observational
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Other Study IDs: INOVA-2023-145
Record Dates: First submitted 2024-02-01; First posted 2024-02-22 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Permanent Sterilization; Pregnancy Related
Keywords: Sterilization, salpingectomy, cesarean delivery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Complete salpingectomy using a hand-held bipolar energy instrument
  Interventions: Other: Hand-held bipolar energy instrument
- Complete salpingectomy using traditional suture ligation
  Interventions: Other: Traditional suture ligation

INTERVENTIONS:
Other: Hand-held bipolar energy instrument — A bipolar energy instrument is used for complete salpingectomy at the time of cesarean delivery.
  Groups: Complete salpingectomy using a hand-held bipolar energy instrument
Other: Traditional suture ligation — Traditional suture ligation technique is used for complete salpingectomy at the time of cesarean delivery.
  Groups: Complete salpingectomy using traditional suture ligation

SUMMARY:
One in three women of reproductive age utilize tubal sterilization for contraception, and sterilization is often requested at time of cesarean delivery. Complete salpingectomy for the purpose of permanent sterilization at the time of cesarean birth is increasingly being performed worldwide.

A preferred complete salpingectomy technique for the purpose of sterilization at the time of cesarean delivery has not emerged in current practice. The objective is to compare short-term clinical outcomes and cost of salpingectomy using a hand-held bipolar energy instrument with those of traditional suture ligation. This retrospective cohort study will be conducted from 2017-2023 at a single tertiary care hospital. The investigators hypothesize that bipolar energy instrument use will not significantly improve clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* request for permanent sterilization at the time of cesarean delivery
* 24 weeks' gestation or beyond
* 21 years old or older
* Medicaid sterilization consent per Virginia Department of Medical Assistance Services regulations (if Medicaid recipient).

Exclusion Criteria:

* vaginal delivery
* history of prior adnexal surgery (such as prior bilateral tubal ligation or unilateral salpingectomy oophorectomy)
* placenta accreta spectrum
* placenta previa
* history of bleeding diathesis.

Min Age: 21 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients aged 21 years or older undergoing permanent sterilization at the time of cesarean delivery at 24 weeks' gestation or beyond, 21 years old and older
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin levels on postoperative day one | preoperatively and one day after surgery
  Change in hemoglobin levels reported in gram per deciliter on postoperative day one, calculated as the difference between immediate preoperative and postoperative day 1 hemoglobin levels

SECONDARY OUTCOMES:
Completion rate of sterilization | preoperatively and one day after surgery
  Proportion of sterilization procedure completed by postoperative day one
Total procedure estimated blood loss | intraoperatively
  estimated blood loss calculated and documented in milliliters at the end of the procedure
Adjacent organ damage | intraoperatively
  Rate of injury to abdominal/pelvic organs sustained during the procedure
Need for blood transfusion | from day of surgery up to 30 days pospartum
  any need for blood products transfusion intraoperatively through discharge
Total operative time | intraoperatively
  time necessary to complete the surgery from skin incision to end of skin closure
ICU admission | from day of surgery up to 7 days postpartum
  any admission to the intensive care unit for procedure-related complications
Length of hospital stay | from day of surgery up to 6 weeks postpartum
  Duration of hospitalization in days from admission to discharge
Hospital readmission postoperatively | Day of initial dischage through 6 weeks postpartum
  Any admission after initial discharge from the hospital
Reoperation rates | postoperative day 0 through 6 weeks postpartum
  Number of participants who return to the operating room due to initial procedure-related complications
Pain score | from day of surgery up to 7 days postparum
  pain severity measured on a scale of 0 through 10
Surgical site infection | postoperative day 0 through 6 weeks postpartum
  any infection that occurs post-surgery in the abdomen, pelvis, abdominal walls or skin
Cost | intraoperatively
  cost difference between bipolar instrument and suture

CONTACTS AND LOCATIONS:
Overall Officials: Jean W Thermolice, MD, Principal Investigator — Inova Fairfax Medical Campus
Locations (1):
- Inova Fairfax Medical campus, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mandelbaum RS, Matsuzaki S, Sangara RN, Klar M, Matsushima K, Roman LD, Paulson RJ, Wright JD, Matsuo K. Paradigm shift from tubal ligation to opportunistic salpingectomy at cesarean delivery in the United States. Am J Obstet Gynecol. 2021 Oct;225(4):399.e1-399.e32. doi: 10.1016/j.ajog.2021.06.074. Epub 2021 Jun 26. PMID 34181896
- [Background] Venkatesh KK, Clark LH, Stamilio DM. Cost-effectiveness of opportunistic salpingectomy vs tubal ligation at the time of cesarean delivery. Am J Obstet Gynecol. 2019 Jan;220(1):106.e1-106.e10. doi: 10.1016/j.ajog.2018.08.032. Epub 2018 Aug 28. PMID 30170036
- [Background] Subramaniam A, Einerson BD, Blanchard CT, Erickson BK, Szychowski J, Leath CA 3rd, Biggio JR, Huh WK. The cost-effectiveness of opportunistic salpingectomy versus standard tubal ligation at the time of cesarean delivery for ovarian cancer risk reduction. Gynecol Oncol. 2019 Jan;152(1):127-132. doi: 10.1016/j.ygyno.2018.11.009. Epub 2018 Nov 23. PMID 30477808
- [Background] ACOG Committee Opinion No. 774 Summary: Opportunistic Salpingectomy as a Strategy for Epithelial Ovarian Cancer Prevention. Obstet Gynecol. 2019 Apr;133(4):842-843. doi: 10.1097/AOG.0000000000003165. PMID 30913193
- [Background] Society of Gynecologic Oncology. SGO Clinical Practice Statement: Salpingectomy for Ovarian Cancer. 2013. https://www.sgo.org/clinicalpractice/guidelines/sgo-clinical-practice-statement-salpingectomy-for-ovarian-cancer-prevention
- [Background] Walker JL, Powell CB, Chen LM, Carter J, Bae Jump VL, Parker LP, Borowsky ME, Gibb RK. Society of Gynecologic Oncology recommendations for the prevention of ovarian cancer. Cancer. 2015 Jul 1;121(13):2108-20. doi: 10.1002/cncr.29321. Epub 2015 Mar 27. PMID 25820366
- [Background] Nguyen, N. T., Alabaster, A., Simmons, S., Weintraub, M. L. R., & Powell, C. B. (2019). Opportunistic salpingectomy techniques at the time of cesarean delivery: a retrospective cohort study. Journal of Clinical Gynecology and Obstetrics, 8(3), 70-76.
- [Background] Lauterbach R, Gruenwald O, Matanes E, Justman N, Mor O, Vitner D, Avrahami R, Ghanem N, Zipori Y, Weiner Z, Lowenstein L. A randomized controlled trial of 2 techniques of salpingectomy during cesarean delivery. Am J Obstet Gynecol MFM. 2022 Nov;4(6):100690. doi: 10.1016/j.ajogmf.2022.100690. Epub 2022 Jul 16. PMID 35843545
- [Result] Chan LM, Westhoff CL. Tubal sterilization trends in the United States. Fertil Steril. 2010 Jun;94(1):1-6. doi: 10.1016/j.fertnstert.2010.03.029. PMID 20497790